CLINICAL TRIAL: NCT02356380
Title: The Effects of Thoracic Spine Mobilizations in Individuals With Neck Pain.
Acronym: THSPMOBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chatham University (Other)
Responsible Party: Principal Investigator, Steve Karas, Assistant Professor, Chatham University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChathamU
Record Dates: First submitted 2015-02-02; First posted 2015-02-05 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobilization (Experimental): Group One: Mobilization Group: this group will receive grade 1,2,3,or 4 mobilization in prone based on the PT's clinical judgement. The treatment parameters will be recorded.
  Group Two: Grade 3-4 mobilization group: this group will receive a grade 3-4 mobilization, for 30 seconds form the first through sixth thoracic vertebrae.
  Interventions: Other: Mobilization Type

INTERVENTIONS:
Other: Mobilization Type — Group One: Mobilization Group: this group will receive grade 1,2,3,or 4 mobilization in prone based on the PT's clinical judgement. The treatment parameters will be recorded.
  Group Two: Grade 3-4 mobilization group: this group will receive a grade 3-4 mobilization, for 30 seconds form the first through sixth thoracic vertebrae.

SUMMARY:
To determine the affects of Physical Therapists clinical reasoning using thoracic spine mobilization for neck pain compared to a standard protocol.

DETAILED DESCRIPTION:
The purpose of this research is to compare the effects of two commonly used, safe, thoracic spine treatments: grade 1-4 as performed by Cleland et. al. and grade 1-4 mobilization to the thoracic spine as selected by the Physical Therapist for cervical spine pain. The immediate effects of thoracic spine mobilization have been shown to facilitate greater range of motion increases in the cervical spine and greater pain decreases within a treatment session and on follow-up visits. There is no research utilizing pain threshold perception as an objective outcome of these treatments. Only one study compared the two treatment techniques and concluded that future research should be completed which includes manual therapy for the thoracic spine. (Cleland 2007) If the PT identifies an appropriate patient they will ask if they are interested in being a research subject. The Physical Theapist recruiting subjects all have completed their Doctor of Physical Therapy Degree and have advanced training in manual Physical Therapy. The techniques employed are considered standard practice and are defined as entry level skills by the Comission of Accredicdation of Physical Therapy Programs. These techniques are typically taught in DPT degree programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Neck Pain
* Ages 18 - 60

Exclusion Criteria:

* Red flags: leg weakness, night pain, history of cancer, upper motor neuron signs, infection, tumors, osteoporosis, fracture (Boissonnault, 2011) (Cleland, 2004), cervical stenosis, CNS involvement, signs consistent with nerve root compression, previous surgery, pending legal action

The inclusion and exclusion above represent a conservative approach based on combining criteria of recent studies in published review articles. (Cross, 2011; Walser, 2009

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Neck Pain | 2 weeks
  0-10 scale
Neck Disability Index | 2 weeks
  Assessment of function of neck using a valid and reliable written tool.
Global Rating of Change | 2 weeks
  A written scale assessing overall improvement

CONTACTS AND LOCATIONS:
Locations (1):
- Chatham University, Pittsburgh, Pennsylvania, United States